CLINICAL TRIAL: NCT01941862
Title: Development and Evaluation of a Brief, Suicide Prevention Intervention Targeting Anxiety and Mood Vulnerabilities
Brief Title: Depression and Anxiety Reduction Treatment for Suicide
Acronym: DARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-10-2-0181
Record Dates: First submitted 2013-07-20; First posted 2013-09-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Anxiety; Depression; Suicide
Keywords: computerized intervention; cognitive bias modification; anxiety; mood; perceived burdensomeness; thwarted belongingness; suicide; post-traumatic stress disorder
MeSH Terms: conditions — Anxiety Disorders; Depression; Suicide; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Anxiety Risk Reduction (Experimental): The anxiety risk reduction condition will be a combination of psychoeducation plus Cognitive Bias Modification (CBM-I) for anxiety sensitivity (AS). The psychoeducational component will focus on the nature of stress and its effect on the body. Interoceptive exposure (IE) exercises, designed to correct the conditioned fear to these bodily sensations, will be explained and practiced.
  Interventions: Behavioral: Psychoeducation and Cognitive Bias Modification
- Mood Risk Reduction (Experimental): The mood risk reduction condition will be a combination of psychoeducation plus Cognitive Bias Modification (CBM-I) for perceived burdensomeness and thwarted belongingness. The psychoeducational component will focus on dispelling myths related to burdensomeness and belongingness and describe their role in the development of mood symptoms.
  Interventions: Behavioral: Psychoeducation and Cognitive Bias Modification
- Combined Risk Reduction (Experimental): The combined intervention will involve all of the interventions in the anxiety and mood risk reduction conditions and thus will not be matched for length.
  Interventions: Behavioral: Psychoeducation and Cognitive Bias Modification
- Repeated Contact Control (No Intervention): Participants assigned to the repeated contact group will be assigned a "personal" study coordinator. The coordinator will contact them at specific intervals during the study. The rationale for these contacts will be provided (e.g., checking in on their status and helping to administer some brief measures). During the three weeks (corresponding to treatment session intervals for those in one of the active treatment conditions), the study coordinator will contact the participant once per week for a brief phone check in where suicide risk will be evaluated. Participants in the control group will also meet with their study coordinator during each of the scheduled follow-up visits.

INTERVENTIONS:
Behavioral: Psychoeducation and Cognitive Bias Modification
  Arms: Anxiety Risk Reduction; Combined Risk Reduction; Mood Risk Reduction

SUMMARY:
The purpose of this study is to test the effectiveness and usability of multiple computer-based treatments for mood and anxiety relevant risk factors. The target of the treatment is related to cognitive stress, which has been shown to be associated with a variety of negative mental health outcomes such as Post-Traumatic Stress Disorder, suicidal ideation, and substance use disorders.

DETAILED DESCRIPTION:
DARTS is a newly developed computerized treatment targeting specific risk factors associated with suicide, mood, and anxiety symptoms. Eligible individuals will be randomized to one of several conditions. In all conditions, participants will complete various self-report questionnaires and a neurophysiology assessment that involves an EEG. Some participants will also be asked to complete four additional EEG assessments. In addition, all participants will be asked to complete a 1, 3, and 6-month follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* At or above community sample mean on ASI-3
* At or above community sample mean on INQ-R
* English speakers
* 18 years of age or older

Exclusion Criteria:

* Significant medical illness
* Current substance dependence
* Current or past psychotic-spectrum disorders
* Uncontrolled bipolar disorder
* Serious suicidal intent that warranted immediate treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Interpersonal Needs Questionnaire (INQ) | Month 6 follow-up
  The INQ is a 15-item self-report measure of the constructs of thwarted belongingness and perceived burdensomeness as defined by the Interpersonal Theory of Suicide. Van Orden et al. report high internal consistency coefficients for the thwarted belongingness (α=.85) and perceived burdensomeness subscales (α=.89). In support of construct validity, both subscales were found to prospectively predict suicidal ideation.

SECONDARY OUTCOMES:
Anxiety Sensitivity Index-3 (ASI-3) | Month 6 follow-up
  The ASI-3 is an 18-item self-report measure of anxiety sensitivity (AS). This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the original ASI provides. Each subfactor is represented by six items. The measure has shown good psychometric properties.

OTHER OUTCOMES:
Beck Suicide Scale (BSS) | Month 6 follow-up
  The BSS is a 21-item widely used self-report measure assessing a broad spectrum of behaviors and attitudes related to suicide risk, including suicidal ideation and past suicide attempts. It has demonstrated strong reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Santopetro NJ, Thompson B, Albanese B, Brush CJ, Schmidt NB. Depression Remission Over Six Months Characterized by Elevated Target-Locked P300 ERP Component: Prospective Evidence Employing an Affective Visual Oddball Task. Psychophysiology. 2025 May;62(5):e70067. doi: 10.1111/psyp.70067. PMID 40345151
- [Derived] Capron DW, Allan NP, Schmidt NB. The Depression Sensitivity Index: Initial Development and Tests of Convergent and Construct Validity. J Affect Disord. 2021 May 15;287:417-426. doi: 10.1016/j.jad.2021.03.051. Epub 2021 Mar 31. PMID 33839487
- [Derived] Short NA, Stentz L, Raines AM, Boffa JW, Schmidt NB. Intervening on Thwarted Belongingness and Perceived Burdensomeness to Reduce Suicidality Among Veterans: Subanalyses From a Randomized Controlled Trial. Behav Ther. 2019 Sep;50(5):886-897. doi: 10.1016/j.beth.2019.01.004. Epub 2019 Jan 24. PMID 31422845
- [Derived] Macatee RJ, Albanese BJ, Clancy K, Allan NP, Bernat EM, Cougle JR, Schmidt NB. Distress intolerance modulation of neurophysiological markers of cognitive control during a complex go/no-go task. J Abnorm Psychol. 2018 Jan;127(1):12-29. doi: 10.1037/abn0000323. PMID 29369665
- [Derived] Short NA, Boffa JW, Norr AM, Albanese BJ, Allan NP, Schmidt NB. Randomized Clinical Trial Investigating the Effects of an Anxiety Sensitivity Intervention on Posttraumatic Stress Symptoms: A Replication and Extension. J Trauma Stress. 2017 Jun;30(3):296-303. doi: 10.1002/jts.22194. Epub 2017 Jun 6. PMID 28585746